CLINICAL TRIAL: NCT02196974
Title: Bronchoscopic Approach to the Peripheral Lung Nodule - Endobronchial Ultrasound, Electromagnetic Navigation and Cryobiopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Paul MacEachern, Clinical Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24185
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Lung Nodules
Keywords: bronchoscopy; lung nodule; diagnosis; cryobiopsy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cryobiopsy (Experimental)
  Interventions: Procedure: cryobiopsy

INTERVENTIONS:
Procedure: cryobiopsy

SUMMARY:
In patients with peripheral lung nodules, what is the additional diagnostic yield of biopsies obtained with flexible cryoprobes compared to standard techniques? For patients with peripheral nodules, we hypothesize use of the cryoprobe will allow larger samples of tissue to be obtained and therefore, will increase the diagnostic yield over conventional techniques

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >18 years 2. Lung nodule (s) identified on CT scan 3. Clinical decision to obtain tissue biopsy of lung lesion 4. CT guided biopsy not preferred technique

  * Previous negative CT guided biopsy
  * Technically difficult nodule location
  * Perceived high risk of pneumothorax or other complications

Exclusion Criteria:

* 1. Lack of informed consent 2. Nodule less than 1 cm or greater than 6 cm long axis 3. Significant mediastinal adenopathy. 4. No suspected sites of disease outside the thorax amenable to biopsy 5. Evidence of endobronchial abnormality on chest CT 6. Medical contraindication to bronchoscopy 7. Patients with lesions highly suspicious for lung cancer, potentially resectable with lobar or lesser resection and without significantly increased operative risk factors will not be entered into this study prior to surgical evaluation.

  8. Uncontrolled or irreversible coagulopathy
  * platelets <100
  * INR >1.3
  * Use of clopidogrel in the 7 days prior to bronchoscopy 9. Confirmed or suspected pregnancy 10. Clinically unable to tolerate a pneumothorax or single-lung ventilation 11. Pacemaker or implanted cardiac defibrillator if it is felt that ENB is needed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
incremental diagnostic yield of cryobiopsy over the standard specimens | 1 year after completion of recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada